CLINICAL TRIAL: NCT01819727
Title: A Phase 3, Open-Label, Randomized, Multi-Center Study to Assess the Safety & Tolerability of an Induction, Titration, and Maintenance Dose Regimen of BMN 165 Self Administered by Adults With PKU Not Previously Treated With BMN 165
Brief Title: An Open-Label Phase 3 Study of BMN 165 for Adults With PKU Not Previously Treated w/ BMN 165
Acronym: Prism301
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 165-301; Prism301 (Other: Phase 3 "brand" name)
Record Dates: First submitted 2013-03-18; First posted 2013-03-28 (Estimated); Results first posted 2018-09-10 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Phenylketonuria
Keywords: PKU; PEG-PAL; BioMarin; rAv-PAL PEG; BMN 165; open label; Prism301; Pegvaliase
MeSH Terms: conditions — Phenylketonurias | interventions — pegvaliase

STUDY DESIGN:
Masking Description: All subjects receive Study Drug. Subjects will be randomized (1:1) to titrate up to one of two dose regimens: 20 mg/day or 40 mg/day.Eligible subjects will be randomized 1:1 using an IWRS to titrate to one of two dose regimens:
  20 mg/day or 40 mg/day. The randomization will be stratified by blood Phe levels of 600 to 900 µmol/L and >900 µmol/ using the last available blood Phe concentration prior to Day 1 of the study.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BMN 165, 20mg/day (Active Comparator): Subjects who meet the eligibility criteria will be randomized 1:1 to titrate to one of two dose regimens: 20 mg/day or 40 mg/day. The randomization will be stratified by the last available blood Phe concentration prior to Day 1 (600 to 900 μmol/L and > 900 μmol/L).
  Interventions: Drug: BMN 165
- BMN 165, 40mg/day (Active Comparator): Subjects who meet the eligibility criteria will be randomized 1:1 to titrate to one of two dose regimens: 20 mg/day or 40 mg/day. The randomization will be stratified by the last available blood Phe concentration prior to Day 1 (600 to 900 μmol/L and > 900 μmol/L).
  Interventions: Drug: BMN 165

INTERVENTIONS:
Drug: BMN 165 — After informed consent, eligible subjects will be randomized (1:1) to titrate up to one of two dose regimens: 20 mg/day or 40 mg/day. All subjects will initiate IP at a fixed-dose of 2.5 mg/week for 4 weeks (Induction). After the Induction Period, subjects will enter the Titration Period (Weeks 5 up to 34) where they will increase their weekly BMN 165 dose to a daily dose regimen of 20 mg/day or 40 mg/day. The Titration Period will be individualized to each subject based on a minimum of 6 weeks (the amount of time it takes to reach a dose regimen of 20 mg/day with no dose interruptions) and up to 30 weeks (accounts for dose reduction or interruption due to AEs). Subjects will stop titration once they have achieved either the 20 mg/day or 40 mg/day dose regimen. The majority of subjects will maintain the 20 or 40 mg/day dose regimen for at least an additional 2 weeks until a minimum of approximately 26 weeks or a maximum of 36 weeks in the study.
  Other Names: rAvPAL-PEG; Pegvaliase

SUMMARY:
The BMN 165 clinical development program has been designed to demonstrate the safety and efficacy of BMN 165 in reducing blood Phe concentrations in patients 18 to 70 years old with hyperphenylalaninemia due to PKU. Study BMN 165-301 is a Phase 3, open-label, randomized study designed to further characterize the safety of BMN 165 during two induction, titration, and maintenance dose regimens in adults with PKU who have not had previous exposure to BMN 165 (naive). Subjects will be randomized (1:1) to titrate up to one of two dose regimens. Other key features of this study are the dose regimens chosen for induction and titration; the study duration; self administration of study drug; and the chosen tertiary objectives.

DETAILED DESCRIPTION:
Primary and Secondary Outcomes:

The primary objective of the study is the following:

* To characterize the safety and tolerability during induction, titration, and maintenance dosing in BMN 165-naïve subjects who self administer BMN 165 at dose levels of 20 mg/day and 40 mg/day

The secondary objective of the study is the following:

* To evaluate blood Phe concentration during induction, titration, and maintenance dosing in BMN 165-naïve subjects who self administer BMN 165 at dose levels of 20 mg/day and 40 mg/day

The tertiary objectives of the study are the following:

* Percentage of daily recommended intake for age of natural protein intake
* Dietary protein intake from medical food and intact food
* The ADHD-RS score (-Investigator Rated; inattentive subscale score, total score, and hyperactivity/impulsivity subscale score)
* POMS scores (-Observer Rated and -Subject Rated)
* Trough plasma concentrations of BMN 165

Primary Analysis:

All AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). The incidence of AEs will be summarized by system organ class, preferred term, relationship to study drug, and severity for the subjects who are randomized to the 40 mg/day dose, the 20 mg/day dose, and overall. A by-subject listing will be provided for those subjects who experience an SAE, including death, or experience an AE associated with early withdrawal from the study or study drug. Hypersensitivity AEs and AEs that result in dosing interruption or dose reduction are of interest, and the percentage of subjects who report these AEs will be presented.

Clinical laboratory data will be summarized by the type of laboratory test for the subjects who are randomized to the 40 mg/day dose, the 20 mg /day dose, and overall. Frequency and percentage of subjects who experience abnormal (ie, outside of reference range) and/or clinically significant abnormalities after study drug administration will be presented for each clinical laboratory test. For each clinical laboratory test, descriptive statistics will be provided for baseline and all subsequent post-baseline visits. Changes from baseline to the post-baseline visits will also be provided. Descriptive statistics, including clinically significant changes from baseline, of vital signs, physical examination results, ECG test results, and immunogenicity test results will also be provided in a similar manner. Additionally, antibodies and titers will be summarized at the scheduled time point.

Detailed statistical methods will be provided in the Statistical Analysis Plan (SAP).

Secondary Analysis:

The secondary efficacy endpoint is change from baseline to end of study in blood Phe concentration.

Baseline is defined as the average of blood Phe concentrations collected prior to dosing at the Screening Visit and on Day 1.

The primary analysis method for the secondary endpoint will use a repeated measures model, with change from baseline Phe as the dependent variable and dose (40 mg/day or 20 mg/day), study week, and baseline Phe as independent variables.

A responder analysis will be presented as a cumulative distribution function. The percentage of subjects with blood Phe concentration below "X" umol/L at the end of the study will be plotted and summarized for various "X" as a cumulative distribution function for each of the 2 doses and overall.

Detailed statistical methods will be provided in the SAP.

Tertiary Analyses:

The statistical analysis method for tertiary endpoints (protein intake; the ADHD-RS IV score) will be descriptive. More details regarding the analysis methods for the tertiary endpoints will be provided in the SAP.

Trough plasma concentrations of BMN 165 will be evaluated.

DMC The Data Monitoring Committee (DMC) will act in an advisory capacity to

BioMarin to monitor subject safety and the efficacy of BMN 165 in subjects who participate in Study BMN 165-301 .The DMC responsibilities may include the following:

* Review the study protocol, informed consent and assent documents, and plans for data monitoring
* Evaluate the progress of the trial; study data quality; timeliness; subject recruitment, accrual and retention; subjects' risk versus benefit; and other factors that could affect the study outcome
* Consider relevant information that may have an effect on the safety of the participants or the ethics of the study
* Protect the safety of the study participants in accordance with the stopping rules as defined in study protocol
* Make recommendations to BioMarin concerning continuation or termination of the study or other modifications of the study based on their observations
* If appropriate, conduct interim analysis of safety and efficacy

ELIGIBILITY:
INCLUSION CRITERIA

Individuals eligible to participate in this study must meet all of the following criteria:

* A current diagnosis of PKU with the following:

  * Current blood Phe concentration >600 µmol/L at screening and
  * Average blood Phe concentration of >600 µmol/L over the past 6 months (per available data)
* Have no previous exposure to BMN 165
* Are ≥18 and ≤70 years of age at the time of screening

  * Subjects who are < 18 years of age but are already enrolled into the study may continue to participate
* If taking Kuvan, have a treatment end date ≥14 days prior to Day 1 (ie, first dose of BMN 165)
* Are willing and able to provide written, signed informed consent after the nature of the study has been explained and prior to any research-related procedures
* Are willing and able to comply with all study procedures
* Has identified a person who is ≥ 18 years of age who has the neurocognitive and linguistic capacities to comprehend and complete the POMS-Observer-rated scale
* Has identified a competent person or persons who are ≥ 18 years of age who can observe the subject during study drug administration and for a minimum of 1 hour following administration until dose titration has completed and if needed upon return to dosing after an AE and per investigator determination.

  * A home healthcare nurse may perform the study drug observations.
* For females of childbearing potential, must have a negative pregnancy test at screening and be willing to have additional pregnancy tests during the study. (Females are considered not of childbearing potential if they have been in menopause for at least 2 years, have had a tubal ligation at least 1 year prior to screening, or have had a total hysterectomy.)
* If sexually active, must be willing to use 2 acceptable methods of contraception while participating in the study and 4 weeks after the study.

  * Males post vasectomy 2 years with no known pregnancies for at least 2 years do not need to use any other forms of birth control during the study.
  * Females who have been in menopause for at least 2 years, have had a tubal ligation at least 1 year prior to screening, or have had a total hysterectomy do not need to use any other forms of contraception during the study.
* Have received documented approval from a study dietician confirming that the subject is capable of maintaining their diet in accordance with dietary information presented in the protocol.
* Have neurocognitive and linguistic capacities to comprehend and answer investigator's prompts for the ADHD RS- Investigator rated instrument and to complete the POMS-Subject rated scale.
* If applicable, maintained stable dose of medication for attention deficit hyperactivity disorder (ADHD), depression, anxiety, or other psychiatric disorder for ≥8 weeks prior to enrollment and willing to maintain stable dose throughout study unless a change is medically indicated.
* Are in generally good health, as evidenced by physical examination, clinical laboratory evaluations and ECG tests performed at screening

EXCLUSION CRITERIA

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

* Use of any investigational product or investigational medical device within 30 days prior to screening or requirement for any investigational agent prior to completion of all scheduled study assessments.
* Use of any medication that is intended to treat PKU (except Kuvan), including the use of large neutral amino acids, within 2 days prior to administration of study drug Day 1 (first dose of BMN 165). Note: Kuvan treatment must be stopped ≥14 days before Day 1
* Use or planned use of any injectable drugs containing PEG (other than BMN 165), including medroxyprogesterone injection, within 3 months prior to screening and during study participation
* Known hypersensitivity to any components of BMN 165
* Current use of levodopa
* A positive test for HIV antibody, hepatitis B surface antigen, or hepatitis C antibody
* A history of organ transplantation or on chronic immunosuppressive therapy
* A history of substance abuse (as defined by the Diagnostic and Statistical Manual of Mental Disorders [DSM IV]) in the past 12 months or current alcohol or drug abuse
* Current participation in the Kuvan registry study (PKU Demographics, Outcomes and Safety [PKUDOS]). Patients may discontinue the PKUDOS registry trial to allow enrollment in this study
* Pregnant or breastfeeding at screening or planning to become pregnant (self or partner) or breastfeed at any time during the study
* Concurrent disease or condition that would interfere with study participation or safety (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease)
* Major surgery planned during the study period
* Any condition that, in the view of the investigator, places the subject at high risk of poor treatment compliance or terminating early from the study
* Alanine aminotransferase (ALT) concentration ≥2 times the upper limit of normal
* Creatinine >1.5 times the upper limit of normal.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2013-05; Primary Completion 2015-11-25 (Actual); Study Completion 2015-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Merilainen, MD, Study Director — BioMarin Pharmaceutical
Locations (31):
- United States (31):
  - University of California, Altman Clinical and Translational Research Institute, La Jolla, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - The Children's Hospital Colorado, Aurora, Colorado
  - University of Florida Clinical Research Center, Gainesville, Florida
  - University of Miami Health System, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Emory Universty, Decatur, Georgia
  - Ann and Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Children's Hospital, Indianapolis, Indiana
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Weisskopf Child Evaluation Center / University of Louisville, Louisville, Kentucky
  - Boston Children's Hospital, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - University of Missouri, Columbia, Missouri
  - Washington University Center for Applied Research Sciences, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cooper Health Systems, Camden, New Jersey
  - Atlantic Health System - Morristown Medical Center, Morristown, New Jersey
  - Albany Medical College, Albany, New York
  - Icahn School of Medicine at Mount Sinai Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - University Hospital Cleveland, Case Medical Center, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Science at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Washington Medical Center, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bilder DA, Arnold GL, Dimmock D, Grant ML, Janzen D, Longo N, Nguyen-Driver M, Jurecki E, Merilainen M, Amato G, Waisbren S. Improved attention linked to sustained phenylalanine reduction in adults with early-treated phenylketonuria. Am J Med Genet A. 2022 Mar;188(3):768-778. doi: 10.1002/ajmg.a.62574. Epub 2021 Nov 26. PMID 34826353
- See also: Biomarin Pharmaceutical website — http://www.bmrn.com
- See also: BioMarin sponsored PKU educational/community website — http://www.pku.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- BMN 165, 20mg/Day; BMN 165, 40mg/Day: Subjects who meet the eligibility criteria will be randomized 1:1 to titrate to one of two dose regimens: 20 or 40 mg/day. Randomization will be stratified by the last available blood Phe concentration prior to Day 1 (600-900 μmol/L and > 900 μmol/L). All subjects will initiate IP at a fixed-dose of 2.5 mg/week for 4 weeks (Induction). After the IP, subjects will enter the Titration Period (Weeks 5 up to 34) where they will increase their weekly dose to a daily dose regimen of 20 or 40 mg/day. The Titration Period will be individualized to each subject based on a minimum of 6 weeks (the amount of time it takes to reach a dose regimen of 20 mg/day with no dose interruptions) and up to 30 weeks (accounts for dose reduction or interruption due to AEs). Subjects will stop titration once they have achieved either the 20 or 40 mg/day dose regimen. The majority of subjects will maintain the 20 or 40 mg/day dose regimen for at least an additional 2 weeks until 26 weeks-36 weeks in the study.
Period: Overall Study
Arm/Group | BMN 165, 20mg/Day | BMN 165, 40mg/Day
Started | 131 | 130
Completed | 111 | 102
Not Completed | 20 | 28
Not completed — Adverse Event | 8 | 9
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 3 | 2
Not completed — Pregnancy | 1 | 0
Not completed — Protocol Violation | 0 | 2
Not completed — Study Terminated by Sponsor | 0 | 1
Not completed — Withdrawal by Subject | 6 | 11
Not completed — Unable to demostrate ability self-inject | 0 | 1
Not completed — Quit due to lack of health benifits | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMN 165, 20mg/Day | BMN 165, 40mg/Day | Total
Number analyzed (Participants) | 131 | 130 | 261
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.2 (8.63) | 28.1 (8.77) | 29.2 (8.75)
Age, Customized [Count of Participants; unit: Participants]
  16 - <18 years | 5 | 6 | 11
  18 - <66 years | 126 | 124 | 250
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 68 | 130
  Male | 69 | 62 | 131
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 7
  Not Hispanic or Latino | 125 | 128 | 253
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 130 | 124 | 254
  Other | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 131 | 130 | 261

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hypersensitivity Adverse Reaction
Description: Hypersensitivity AEs will be identified in two ways:
  * Broad Algorithmic anaphylactic reaction Standardized MedDRA Queries (SMQ)
  * Modified Hypersensitivity SMQ to include above additional preferred terms
Time Frame: baseline and 36 weeks
Population: The safety population will consist of all subjects who receive any pegvaliase throughout the study duration. The safety population will be analyzed according to the treatment assignment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | BMN 165, 20mg/Day | BMN 165, 40mg/Day
Number analyzed (Participants) | 131 | 130
Participants | 111 | 119

2. Secondary Outcome: Blood Phenylalanine Concentration
Description: Plasma phenylalanine (Phe) concentration
Time Frame: baseline and 36 weeks
Population: The intent-to-treat (ITT) population will consist of all subjects who are randomized to study treatment whether or not treatment was received.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | BMN 165, 20mg/Day | BMN 165, 40mg/Day
Number analyzed (Participants) | 131 | 130
umol/L
  Baseline | 1241.0 (389.70) | 1224.4 (384.28)
  Week 36 | 868.4 (501.78) | 624.4 (530.58)

3. Other Pre Specified Outcome: Dietary Phenylalanine
Description: All patients will complete a 3-day diet diary in order to assess dietary phenylalanine intake.
Time Frame: baseline and 36 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | BMN 165, 20mg/Day | BMN 165, 40mg/Day
Number analyzed (Participants) | 131 | 130
mg
  Baseline | 1750.8 (1168.91) | 1647.9 (1222.68)
  Week 36 | 1851.8 (1145.06) | 2057.9 (1448.21)

ADVERSE EVENTS:
Time Frame: Week 0- Week 36
Arm/Group | BMN 165, 20mg/Day | BMN 165, 40mg/Day
All-Cause Mortality (participants affected / at risk) | 1/131 | 0/130
Serious Adverse Events (participants affected / at risk) | 7/131 | 19/130
Other Adverse Events (participants affected / at risk) | 130/131 | 129/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 165, 20mg/Day (N=131) | BMN 165, 40mg/Day (N=130)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Electrocution (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Puncture site haemorrhage (General disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 6 (6)
Anaphylactoid reaction (Immune system disorders) | 0 (0) | 2 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 3 (3)
Serum sickness (Immune system disorders) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 165, 20mg/Day (N=131) | BMN 165, 40mg/Day (N=130)
Lymphadenopathy (Blood and lymphatic system disorders) | 12 (21) | 10 (18)
Abdominal discomfort (Gastrointestinal disorders) | 11 (13) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 9 (10) | 5 (8)
Abdominal pain upper (Gastrointestinal disorders) | 10 (13) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 13 (16) | 11 (13)
Dyspepsia (Gastrointestinal disorders) | 8 (13) | 9 (11)
Nausea (Gastrointestinal disorders) | 29 (38) | 22 (28)
Vomiting (Gastrointestinal disorders) | 21 (33) | 16 (20)
Chills (General disorders) | 15 (22) | 9 (13)
Fatigue (General disorders) | 21 (58) | 13 (27)
Injection site bruising (General disorders) | 24 (65) | 26 (44)
Injection site erythema (General disorders) | 57 (323) | 61 (210)
Injection site haemorrhage (General disorders) | 7 (9) | 4 (6)
Injection site oedema (General disorders) | 0 (0) | 7 (112)
Injection site pain (General disorders) | 27 (63) | 29 (55)
Injection site pruritus (General disorders) | 29 (87) | 36 (119)
Injection site rash (General disorders) | 22 (96) | 28 (66)
Injection site reaction (General disorders) | 80 (700) | 68 (495)
Injection site swelling (General disorders) | 23 (70) | 20 (45)
Injection site urticaria (General disorders) | 10 (27) | 14 (25)
Oedema peripheral (General disorders) | 6 (7) | 9 (22)
Pain (General disorders) | 22 (31) | 7 (11)
Pyrexia (General disorders) | 26 (43) | 8 (13)
Hypersensitivity (Immune system disorders) | 4 (4) | 7 (7)
Nasopharyngitis (Infections and infestations) | 24 (33) | 25 (29)
Sinusitis (Infections and infestations) | 9 (10) | 13 (13)
Upper respiratory tract infection (Infections and infestations) | 22 (27) | 20 (24)
Contusion (Injury, poisoning and procedural complications) | 17 (26) | 9 (11)
Blood cortisol decreased (Investigations) | 1 (1) | 8 (8)
Blood creatine phosphokinase increased (Investigations) | 7 (7) | 4 (4)
C-reactive protein increased (Investigations) | 12 (16) | 10 (10)
Complement factor C3 decreased (Investigations) | 11 (12) | 7 (7)
Complement factor C4 decreased (Investigations) | 12 (12) | 6 (6)
Red blood cell sedimentation rate increased (Investigations) | 7 (8) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 78 (376) | 92 (350)
Back pain (Musculoskeletal and connective tissue disorders) | 21 (34) | 20 (26)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 8 (9) | 6 (10)
Joint swelling (Musculoskeletal and connective tissue disorders) | 8 (15) | 5 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 (18) | 19 (24)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (18) | 6 (9)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 10 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 (42) | 26 (52)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 8 (9) | 6 (8)
Dizziness (Nervous system disorders) | 20 (24) | 21 (32)
Headache (Nervous system disorders) | 46 (112) | 36 (98)
Anxiety (Psychiatric disorders) | 4 (11) | 10 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 10 (13)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 7 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 22 (23) | 12 (14)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8) | 12 (12)
Erythema (Skin and subcutaneous tissue disorders) | 11 (17) | 12 (28)
Pruritus (Skin and subcutaneous tissue disorders) | 22 (39) | 25 (65)
Rash (Skin and subcutaneous tissue disorders) | 27 (68) | 40 (83)
Rash erythematous (Skin and subcutaneous tissue disorders) | 3 (3) | 8 (17)
Urticaria (Skin and subcutaneous tissue disorders) | 18 (71) | 30 (101)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days